CLINICAL TRIAL: NCT06444607
Title: HEPHESTOS - Hereditary Pheochromocytoma Assessment of Tumour Immunologies
Brief Title: Hereditary Pheochromocytoma Assessment of Tumour Immunologies
Acronym: HEPHESTOS
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 115703
Record Dates: First submitted 2024-05-22; First posted 2024-06-05 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-05

CONDITIONS: Pheochromocytoma; Paraganglioma
Keywords: Pheochromocytoma; Paraganglioma; Tumor microenvironment; Innate immunity
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Serum, plasma, and white blood cells from participating patients, obtained from whole blood during routine care.
  Histological samples from PPGL tissue after planned surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with hereditary PPGL: Blood will be collected prior and after surgery for their pheochromocytoma/paraganglioma (as planned by their treating physician). Blood will also be collected prospectively during regular follow-up appointments after 1 year and after 2 years.
  Interventions: Procedure: Venepuncture
- Patients with sporadic PPGL: Blood will be collected prior and after surgery for their pheochromocytoma/paraganglioma (as planned by their treating physician). Blood will also be collected prospectively during regular follow-up appointments after 1 year and after 2 years.
  Interventions: Procedure: Venepuncture
- Asymptomatic carriers of germline mutations predisposing for PPGL: Blood will be collected at inclusion, after 1 year and after 2 years.
  Interventions: Procedure: Venepuncture
- Sex and age matched healthy volunteers: Blood material will be obtained from healthy anonymous donors according to the protocol "Donation of blood by healthy volunteers for experimental in-vitro research" (Human Subjects Review Board approval number: NL84281.091.23).
  Interventions: Procedure: Venepuncture

INTERVENTIONS:
Procedure: Venepuncture — Blood draw in the context of routine patient care, when a venipuncture is already scheduled.
  Groups: Asymptomatic carriers of germline mutations predisposing for PPGL; Patients with hereditary PPGL; Patients with sporadic PPGL
Procedure: Venepuncture — Volunteering for blood draw.
  Groups: Sex and age matched healthy volunteers

SUMMARY:
In this study, the investigators are examining the role of the immune system in pheochromocytoma and paraganglioma. The investigators aim to examine the differences in the immune system between people who have these tumors with and without a hereditary predisposition. The investigators also want to see how the immune system changes during the development of the tumor in people with a hereditary predisposition. Finally, the investigators will compare the data with a control group of people without these tumors. Ultimately, the investigators hope that the results will contribute to the discovery of new immune system-targeted medications for pheochromocytoma and paraganglioma.

DETAILED DESCRIPTION:
Rationale: Pheochromocytoma and Paraganglioma (PPGL) represent rare, catecholamine-secreting tumours (1). Genetic or sporadic mutations, accounting for approximately 70% of cases, significantly contribute to PPGL development, and are categorized into three clusters based on tumour formation mechanisms (2,3). Current treatment options, particularly for advanced or metastatic disease, are limited (4). Understanding the immune system's role and the impact of genetics on tumour immunology in PPGL could unveil crucial insights for therapeutic advancements. Earlier studies emphasized the immunogenic nature of PPGL, highlighting the tumour microenvironment (TME) and circulatory factors as key components (5-7). However, these studies lack specific examination of genotypes' effect on the immune system. This study aims to address this gap in two parts, particularly focusing on differences between genetic clusters.

Objective: To examine the differences in the immune system in PPGL regarding genetics. Part I will examine immune cell composition and response in circulation. Part II will examine immune cell composition in TME.

Study design: Part I will be a partly cross-sectional and partly prospective cohort study. Part II will be a histological study of retrospectively and prospectively collected PPGL samples.

Study population: Part I will include 80 patients with PPGL, 80 carriers of germline mutations predisposing for PPGL, and 40 sex and age matched healthy volunteers. Part II will include histological samples of 80 patients with hereditary disease and 80 patients with sporadic disease.

Main study parameters/endpoints: The main study outcomes are inflammatory molecules and proteins produced by stimulated and unstimulated immune cells from circulation, immune cell composition in histological PPGL samples and in circulation, and their genetic determinants. Secondary outcomes will comprise of transcriptional and epigenetic signature of circulating immune cells, circulating immunomodulating metabolites, trained immunity, and clinical outcomes such as tumour metastasis, survival.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: For patients and mutation carriers, there is no direct benefit in participating in this study. However, by participating, they can contribute to the acquisition of scientific knowledge and the development of new therapeutic targets and novel disease management strategies. Such strategies might benefit patients and mutation carriers in the future if they potentially develop advanced disease. There are no risks associated with the study. There are no interventions other than those related to the regular patient care (venipuncture). Thus, this study is considered to impose a low burden on patients.

ELIGIBILITY:
Inclusion Criteria:

Part I:

* Newly diagnosed patients with PPGL or newly diagnosed patients with (metastatic) PPGL recurrence.
* OR patients with mutations which predispose for the development of PPGL.
* Aged > 18 years.

Part II:

* Confirmed PPGL on pathology.
* Aged > 18 years.

Exclusion Criteria:

* Unable to provide informed consent.
* Active inflammatory or infectious comorbidities.
* Other malignancies which are under active treatment (except for basal cell carcinoma, other in situ carcinomas).
* Using medication interfering with the immune system
* Pregnancy or breastfeeding
* A self-reported alcohol consumption of >21 units per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For part I, the study population will consist of patients who are presenting or are currently under follow-up at the Radboudumc endocrinology department for their PPGL. Eigthy patients will be included with hereditary or sporadic cases of PPGL and an equal number of asymptomatic carriers. The healthy control group will consist of 40 age and sex matched healthy volunteers.
  Part II will include histological samples of 160 patients with PPGL, of which 80 hereditary and 80 sporadic. A large part of the population will overlap between part I and part II, since almost all patients with PPGL undergo surgery for their tumour. These samples will partly be retrospectively collected from the Radboudumc Urology Biobank, where biomaterials from previously treated patients with PPGLs are kept and stored or future scientific research (Human Subjects Review Board approval number: CWOM-9803-0060). The remaining samples will be collected prospectively from patients undergoing surgery for their PPGL.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Immune cell response in circulation, both after stimulation and in an unstimulated state, measured as the concentration of inflammatory molecules and proteins. | Before surgery, 6 weeks after surgery, after 1 year, after 2 years.
  e.g. cytokines
Immune cell composition in histological PPGL specimens and in circulation. | Before surgery, 6 weeks after surgery, after 1 year, after 2 years. Histological specimens will only be obtained during surgery.

SECONDARY OUTCOMES:
Transcriptional and epigenetic signature of circulating immune cells. | Before surgery, 6 weeks after surgery, after 1 year, after 2 years.
Concentration of immunomodulating metabolites in circulation. | Before surgery, 6 weeks after surgery, after 1 year, after 2 years.
  e.g. catecholamines, succinate.
Trained immunity assessment of circulating immune cells. | Before surgery, 6 weeks after surgery, after 1 year, after 2 years.
Tumour recurrence rate | After 1 year, after 2 years.
Metastasis rate | Before surgery, after 1 year, after 2 years.
Survival rate | After 1 year, after 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Margo Dona, PhD, Principal Investigator — Radboud University Medical Center; Henri Timmers, M.D. PhD, Principal Investigator — Radboud University Medical Center; Romana Netea-Maier, M.D. PhD, Principal Investigator — Radboud University Medical Center; Marieke de Laat, M.D. PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available by the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after completion of the study.

REFERENCES:
- [Background] Lenders JW, Eisenhofer G, Mannelli M, Pacak K. Phaeochromocytoma. Lancet. 2005 Aug 20-26;366(9486):665-75. doi: 10.1016/S0140-6736(05)67139-5. PMID 16112304
- [Background] Cascon A, Calsina B, Monteagudo M, Mellid S, Diaz-Talavera A, Curras-Freixes M, Robledo M. Genetic bases of pheochromocytoma and paraganglioma. J Mol Endocrinol. 2023 Jan 24;70(3):e220167. doi: 10.1530/JME-22-0167. Print 2023 Apr 1. PMID 36520714
- [Background] Jhawar S, Arakawa Y, Kumar S, Varghese D, Kim YS, Roper N, Elloumi F, Pommier Y, Pacak K, Del Rivero J. New Insights on the Genetics of Pheochromocytoma and Paraganglioma and Its Clinical Implications. Cancers (Basel). 2022 Jan 25;14(3):594. doi: 10.3390/cancers14030594. PMID 35158861
- [Background] Nolting S, Bechmann N, Taieb D, Beuschlein F, Fassnacht M, Kroiss M, Eisenhofer G, Grossman A, Pacak K. Personalized Management of Pheochromocytoma and Paraganglioma. Endocr Rev. 2022 Mar 9;43(2):199-239. doi: 10.1210/endrev/bnab019. PMID 34147030
- [Background] Tufton N, Hearnden RJ, Berney DM, Drake WM, Parvanta L, Chapple JP, Akker SA. The immune cell infiltrate in the tumour microenvironment of phaeochromocytomas and paragangliomas. Endocr Relat Cancer. 2022 Sep 19;29(11):589-598. doi: 10.1530/ERC-22-0020. Print 2022 Nov 1. PMID 35975974
- [Background] Gao X, Yamazaki Y, Pecori A, Tezuka Y, Ono Y, Omata K, Morimoto R, Nakamura Y, Satoh F, Sasano H. Histopathological Analysis of Tumor Microenvironment and Angiogenesis in Pheochromocytoma. Front Endocrinol (Lausanne). 2020 Nov 10;11:587779. doi: 10.3389/fendo.2020.587779. eCollection 2020. PMID 33244312
- [Background] van der Heijden CDCC, Groh L, Keating ST, Kaffa C, Noz MP, Kersten S, van Herwaarden AE, Hoischen A, Joosten LAB, Timmers HJLM, Netea MG, Riksen NP. Catecholamines Induce Trained Immunity in Monocytes In Vitro and In Vivo. Circ Res. 2020 Jul 3;127(2):269-283. doi: 10.1161/CIRCRESAHA.119.315800. Epub 2020 Apr 3. PMID 32241223